CLINICAL TRIAL: NCT04349319
Title: Development of Three Dimensional Preoperative Planning System for the Osteosynthesis of Distal Humerus Fractures
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Tokyo Medical University (Other)
Responsible Party: Principal Investigator, Yuichi Yoshii, Associate Professor, Department of Orthopaedic Surgery, Tokyo Medical University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 14-21(distal humerus)
Record Dates: First submitted 2020-04-14; First posted 2020-04-16 (Actual); Last update posted 2022-04-27 (Actual); Status verified 2022-04

CONDITIONS: Distal Humerus Fracture
MeSH Terms: conditions — Humeral Fractures, Distal

STUDY DESIGN:
Intervention Model Description: A case control study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Digital preoperative planning (Other): To use digital preoperative planning software
  Interventions: Device: Digital preoperative planning

INTERVENTIONS:
Device: Digital preoperative planning — Before the osteosynthesis of distal humerus fracture, we perform digital preoperative planning.

SUMMARY:
To reproduce anatomical reduction and appropriate implant placement/choices during osteosynthesis for elbow fractures, a 3D preoperative planning system was developed. To assess the utility of 3D digital preoperative planning for the osteosynthesis of distal humerus fractures, the reproducibility of implant reduction shapes and placements in patients with distal humerus fractures will be evaluated.

DETAILED DESCRIPTION:
3D preoperative planning will be applied for four distal humerus fracture cases . The preoperative planning will be performed in order to determine the reduction, placement and choices of implants. After the operation, the accuracy of the reduction and implants choices and placements will be verified. The reductions will be evaluated with an angle between the diaphysis axis and a line connecting the medial epicondyle with the lateral epicondyle and an angle between the diaphysis axis and the articular surface in the coronal plane and distance between the anterior diaphysis and the anterior articular surface in the sagittal plane for the 3D images of distal humerus. The reproducibility will be evaluated by the differences of the parameters between pre- and post-operative images.

ELIGIBILITY:
Inclusion Criteria:

* Distal humerus fracture patients

Exclusion Criteria:

* Patients with a previous history of traumatic injuries to the elbow

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2017-10-01 (Actual); Primary Completion 2024-03 (Estimated); Study Completion 2025-03 (Estimated)

PRIMARY OUTCOMES:
Reduction shape | 1 year
  Reduction shape parameter
Implant placement | 1 year
  Implant placement parametes

CONTACTS AND LOCATIONS:
Locations (1):
- Tokyo Medical University Ibaraki Medical Center, Ami, Ibaraki, Japan

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Yoshii Y, Iwabuchi S, Ikumi A, Kohyama S, Ogawa T, Ishii T. Correlations between 3D preoperative planning and postoperative reduction in the osteosynthesis of distal humeral fractures. J Orthop Surg Res. 2023 Apr 8;18(1):283. doi: 10.1186/s13018-023-03772-y. PMID 37031170